CLINICAL TRIAL: NCT07081425
Title: Effect of Virtual Reality on Surgical Drain Removal: Pain and Anxiety Management
Brief Title: Surgical Drain Removal: Pain and Anxiety Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Refiye Akpolat, Assist. Profesor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123456789
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Pain Management; Pain Management After Surgery; Anxiety After Surgery; Non-Pharmacological Pain Management; Perioperative Nursing; Surgical Drain
Keywords: virtual reality; Pain management; Perioperative Nursing; Surgıcal Drain Removal; Non-pharmacological method
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRG Group (Experimental): The "VR Box V2.0 Virtual Reality Headset 3D" was used as the "virtual reality glasses" used in the study. The device is compatible with Android operating systems and smartphones. It is not a medical device. The headset can be adjusted to the person after being worn. A suitable program that provides 360° VR viewing can be downloaded to a compatible mobile phone and the relevant content can be watched through the program. In this study, the researcher's mobile phone was used for VRG. Previously downloaded 360° videos of at least 5 minutes of nature-forest walks, underwater life and the sky were presented according to the patients' preferences. The participant was told that he/she could withdraw from this study at any time without giving any reason.
  Interventions: Device: VRG Group
- Control Group (No Intervention): In routine practice, considering the general condition of patients undergoing bariatric surgery, the drain is removed on the 3rd day. Care was taken to ensure that patients did not receive analgesia for at least 4 hours before the procedure. Before the drain was removed, the patient's NRPS level was assessed and the STAI-I questionnaire was filled out. The drain was removed. After the procedure, the patients' pain perception during the procedure was assessed with the NRPS form. The STAI-I questionnaire was filled out again.

INTERVENTIONS:
Device: VRG Group — Care was taken to ensure that patients did not receive analgesia for at least 4 hours before the procedure. Before drain removal, the patient's NRPS level was assessed, and the STAI-I questionnaire was filled out. The experimental group was given a video to watch before the procedure began, and the use of glasses was explained. VRG was put on the patient, and the drain was removed in the 3rd minute while the video was being watched. After the procedure, the patients' pain perception during the procedure was assessed with the NRPS form. The STAI-I questionnaire was filled out again.
  Other Names: Nonpharmacologıcal Pain Method
  Arms: VRG Group

SUMMARY:
Aim: The aim was to evaluate the effect of using virtual reality glasses (VRG) during surgical drain removal on participants' pain and anxiety levels.

Study design: Randomized controlled trial Material and Method: Sixty participants (30 experimental, 30 control) who underwent obesity surgery at a hospital in Turkey were randomized and included in the study. VRG was used during drain removal in the experimental group. While collecting data, demographic data of the participants was collected with the Personal Information Form. Pain and anxiety levels were measured using the Numerical Rating Pain Scale (NRPS) and the State Anxiety Inventory (STAI-I) before and after the procedure. In the use of VRG, patients watched 360° videos with themes of nature, forests, underwater scenes, and the sky, depending on their preference. The collected data were statistically analyzed.

DETAILED DESCRIPTION:
While virtual reality glasses (VRG) were initially used primarily for gaming and entertainment purposes, today they have begun to find wide application areas in the healthcare sector, especially in education, treatment, rehabilitation, and pain management (Ehizogie Paul Adeghe et al., 2024; Kafes & Ileri, 2025). VR technology has begun to gain an increasingly important place in the healthcare field with its continued development. VR increases the participation of patients in the treatment process and enables the development of more effective and personalized treatment methods (Pillai & Mathew, 2019). VR is an important tool for improving the quality of healthcare by improving treatment processes, supporting the training of healthcare professionals, and enriching the patient experience (Buztepe & Çapik, 2024).

When we look at the areas of use of virtual reality glasses in health, it is used in the treatment of phobias (Isikli et al., 2019) In the rehabilitation processes of pain management (Baghaei et al., 2021; Çevik Aktura et al., 2022; Hoşgör, 2022). Surgical interventions are an important turning point for patients, both physically and psychologically. Factors such as the invasive effects of surgery, damage to body tissues, and removal of foreign objects from the body can cause both physical pain and psychological concerns in patients. Acar (2016) concluded in his research that 77.3% of patients had complaints about pain after the surgical procedure (Acar et al., 2016).

Postoperative pain is a significant complication that negatively affects the patient's physical and psychological health, reduces the quality of life, and prolongs treatment processes. Therefore, effective management of postoperative pain is of great importance for a faster recovery and increased quality of life for the patient (Gürkan et al., 2020). This situation becomes more evident, especially in procedures such as the removal of surgical drains. The pain and anxiety experienced during the removal of drains can negatively affect the recovery process of patients, increase the use of painkillers, cause longer hospital stays, and reduce the overall quality of life (Çevik Aktura et al., 2022) The management of pain and anxiety experienced by patients after surgical interventions is of great importance for both patient comfort and the success of the treatment process. In a study conducted by Vazquez et al. in 2019 with patients undergoing cardiac surgery, the effects of the virtual reality experience were examined. Significant decreases in respiratory rate, mean arterial pressure, pain, and anxiety levels were observed in patients who experienced VR (Agrawal et al., 2019).

VR can help reduce pain by providing a distracting and relaxing environment (Değirmen et al., 2022) . According to the results of a different study, VR stands out as an effective alternative treatment method in acute pain management, especially in young people. VR has been successful in reducing the severity of different types of pain, such as postoperative dressing changes, burn wound dressings, and needlestick and peripheral catheter insertion (Güler et al., 2024; Saleh & Abozed, 2024; Sariköse & Turan, 2024). VR also improved the patient's overall well-being by reducing anxiety, discomfort, and time spent thinking about pain, which negatively impact the patient's overall pain experience (Huang et al., 2022). In cases such as post-operative dressing and drain removal, VR can help reduce pain by distracting the patient and help patients cope with these discomforts by providing relaxing and calming experiences in virtual environments. Since there is no study in the literature on the evaluation of pain and anxiety during drain removal, our study aimed to determine the effect of VR on pain and anxiety levels during drain removal in patients undergoing bariatric surgery.

MATERIAL METHODS Study type: Randomized controlled trial Study sample: This randomized controlled trial was conducted with patients undergoing bariatric surgery in a hospital in Kocaeli, Türkiye. The sample consists of 60 patients who underwent bariatric surgery and met the inclusion criteria for the study (experimental group n=30; control group n=30). The size of the study sample was determined statistically by power analysis. The sample size of each group was calculated as 30 patients for a power of 0.80 and a type I error of 0.05. The calculation was made using the PASS13.0 program (PASS, Kaysville, Utah, USA). Participants were assigned to two groups by computer software using a simple randomization method. During the sample selection of the study, 4 patients who met the inclusion criteria were not included in the study because they did not want to use VRG.

Inclusion Criteria for the Study: Being 18 years of age or older, not having any psychiatric illness, dizziness or vision, hearing, or perception problems, and being willing to participate in the study..

Data collection: Data were collected in the surgical clinic of a private hospital in Kocaeli province between April 2023 and November 2024. "Personal Information Form", "Numerical Rating Pain Scale"(NRPS), and "State Anxiety Inventory (STAI-I)" were used to collect the data.

Personal Information Form: It is a form prepared by researchers that includes questions about demographic data and the surgical history of patients used in similar studies in the literature (Abbasnia et al., 2023; Aslan et al., 2025; Ceyhan et al., 2018; Güler et al., 2024; Sariköse & Turan, 2024). The form included questions about the patient's characteristics (age, gender, place of residence, education level), surgery history, and information about the current surgery (presence of previous surgery, type of current surgery, and time of last analgesia application).

Numerical Rating Pain Scale: It is a one-dimensional scale that determines the severity of pain in adult patients and is frequently used in pain assessment in the literature (Adeboye et al., 2021; Chiarotto et al., 2019; Kim et al., 2022; Özyer & Köse, 2023; Savaş & Kahyaoğlu Süt, 2024). Scores range from 0 to 10, with Zero generally representing "no pain at all," while the upper limit represents "worst possible pain." Higher scores indicate greater pain intensity.

State Anxiety Inventory (STAI-I): The State Anxiety Inventory (STAI-I) determines how an individual feels at a certain moment and under certain conditions. STAI-I was developed by Spielberger in 1970, and its Turkish form was adapted by Öner and Le Compte (1983), and its validity and reliability study was conducted. The scale consists of 20 items. Responses are scored between 1-4. The total score obtained from the scale is between 20-80. A high score indicates a high level of anxiety (Öner & Le Compte, 1983; Spielberger et al., 1970).

Equipment: "VR Box V2.0 Virtual Reality Headset 3D" was used as virtual reality glasses. The device is compatible with Android operating systems and smartphones. The headset can be adjusted to the individual after being attached. A suitable program that allows 360° VR viewing can be downloaded to a compatible mobile phone, and the relevant content can be watched through the program. In this study, the researcher's mobile phone was used for VRG. Previously downloaded 360° videos of at least 5 minutes about nature-forest walks, underwater life, and the sky were presented according to the patients' preferences.

Application: In routine practice, considering the general condition of patients undergoing bariatric surgery, the drain is removed on the 3rd day. Care was taken to ensure that patients did not receive analgesia for at least 4 hours before the procedure. Before drain removal, the patient's NRPS level was assessed, and the STAI-I questionnaire was filled out. The experimental group was given a video to watch before the procedure began, and the use of glasses was explained. VRG was put on the patient, and the drain was removed in the 3rd minute while the video was being watched. After the procedure, the patients' pain perception during the procedure was assessed with the NRPS form. The STAI-I questionnaire was filled out again.

Ethical Aspect of the Study: The study protocol was approved by a university's non-interventional research ethics committee (Date-Decision No:23.03.2023;14/4), and institutional permission was obtained from the hospital administration (Decision No: 14839) where the study was conducted. The ethical principles of the Declaration of Helsinki were followed, and after informing the patients about the study, their verbal and written consents were obtained..

Data Analysis: The data obtained in the study were analyzed using SPSS 25 software. The normal distribution between the variables was analyzed with the 'Shapiro-Wilk', and the homogeneity of the distribution was analyzed with the Levene test. Pearson Correlation analysis was used to determine the correlation between two variables with a normal distribution. Independent Samples t test was used for comparisons between independent groups, and p<0.05 level was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older.
2. Not having any psychiatric illness, dizziness, vision, hearing, or perception problems.
3. Being willing to participate in the study.

Exclusion Criteria:

1. Use of painkillers before the procedure.
2. Use of anxiety medication before the procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (SAAS) | Perioperative/Periprocedural
  Numerical pain rating scale (NPRS) is used to evaluate pain severity. In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).The patient's pain was assessed using the NPRS 15 minutes before surgical drain removal. The drain was removed, and the removal process took 5 minutes. After the procedure, the patient's pain perception during drain removal was re-examined using the NPRS
State Anxiety Scale (STAI TX-I) | Perioperative/Periprocedural
  The State Anxiety Inventory (STAI TX-I) items are answered by selecting one of the following options, depending on the severity of the emotion or behavior: (1) not at all, (2) a little, (3) a lot, or (4) a lot. There are two types of statements on the scale: reversed or direct. Reversed statements express positive emotions, while direct statements express negative emotions. When scoring reversed statements, items with a weight of 1 are converted to 4, and those with a weight of 4 are converted to 1.
  The State Anxiety Inventory has ten reversed statements: items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The reversed and direct statements are added together during scoring. A higher total score indicates a higher anxiety level. The patient was asked to complete the STAI-I form 15 minutes before the drain removal procedure. The drain was removed, and the removal procedure took 5 minutes. After the procedure, the patient's anxiety during drain removal was re-evaluated using STAI-I.

CONTACTS AND LOCATIONS:
Overall Officials: Refiye Akpolat, Principal Investigator — Kocaeli Sağlık ve Teknoloji Üniversitesi, Kocaeli, Türkiye
Locations (1):
- Kocaeli Health and Tecnology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can allow my article to be shared after it is published

REFERENCES:
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210
- [Background] Adeboye A, Hart R, Senapathi SH, Ali N, Holman L, Thomas HW. Assessment of Functional Pain Score by Comparing to Traditional Pain Scores. Cureus. 2021 Aug 3;13(8):e16847. doi: 10.7759/cureus.16847. eCollection 2021 Aug. PMID 34522490
- [Background] Abbasnia F, Aghebati N, Miri HH, Etezadpour M. Effects of Patient Education and Distraction Approaches Using Virtual Reality on Pre-operative Anxiety and Post-operative Pain in Patients Undergoing Laparoscopic Cholecystectomy. Pain Manag Nurs. 2023 Jun;24(3):280-288. doi: 10.1016/j.pmn.2022.12.006. Epub 2023 Jan 17. PMID 36658058
- [Background] Agrawal AK, Robertson S, Litwin L, Tringale E, Treadwell M, Hoppe C, Marsh A. Virtual reality as complementary pain therapy in hospitalized patients with sickle cell disease. Pediatr Blood Cancer. 2019 Feb;66(2):e27525. doi: 10.1002/pbc.27525. Epub 2018 Oct 26. PMID 30362236
- [Background] Baghaei N, Chitale V, Hlasnik A, Stemmet L, Liang HN, Porter R. Virtual Reality for Supporting the Treatment of Depression and Anxiety: Scoping Review. JMIR Ment Health. 2021 Sep 23;8(9):e29681. doi: 10.2196/29681. PMID 34554097
- [Background] Buztepe S, Capik C. The validity and reliability of the emotional consequences of elder abuse scale for Turkish language. BMC Geriatr. 2025 May 23;25(1):369. doi: 10.1186/s12877-025-06026-0. PMID 40410670
- [Background] Kafes, M., & Ileri, Y. Y. (2025). Current status of virtual reality research in healthcare: thematic and bibliometric analysis. Frontiers in Virtual Reality, 6.
- [Background] Adeghe, E. P., Okolo, C. A., & Ojeyinka, O. T. (2024). A review of the integration of virtual reality in healthcare: implications for patient education and treatment outcomes. Int J Sci Technol Res Arch, 6(1), 79-88. https://doi.org/10.53771/ijstra.2024.6.1.0032